CLINICAL TRIAL: NCT04345341
Title: Efficacy of Laparoscopic-assisted Transversus Abdominus Plane (TAP) Block in Minimally Invasive Gynecologic Surgeries: A Prospective, Randomized Control Trial.
Brief Title: Efficacy of Laparoscopic-assisted Transversus Abdominus Plane (TAP) Block Compared to Ultrasound-guided TAP Block in Minimally Invasive Gynecologic Surgeries: A Prospective, Randomized Control Trial.
Acronym: TAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000026422; No NIH funding (Other: 11.07.23)
Record Dates: First submitted 2020-04-01; First posted 2020-04-14 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: the Efficacy of Analgesia of Laparoscopic TAP Block in Minimally Invasive Gynecology Surgeries
Keywords: TAP block , laparoscopy , minimally invasive gynecology
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic assisted TAP block (Active Comparator): Laparoscopic assisted TAP block will be done by surgeon intra-operatively
  Interventions: Drug: TAP block with liposomal bupivacaine and bupivacaine
- no TAP block (No Intervention): no TAP block would be done

INTERVENTIONS:
Drug: TAP block with liposomal bupivacaine and bupivacaine — injecting the mixture of bupivacaine with liposomal bupivacaine in transversus abdominis plane to block the somatic nerves
  Arms: Laparoscopic assisted TAP block

SUMMARY:
We propose a clinical trial to determine the efficacy of Laparoscopic Transversus Abdominis Plane (LA-TAP) performed intraoperatively compared with usual postoperative analgesia without LA-TAP block. We hypothesise that there will be a decrease in postoperative opioid utilization and in pain scores for patients randomized to receive the LA-TAP block verses those who do not. We expect that patients will opt to take less break through opioid medication in the LA-TAP block group versus the no TAP block group.

Investigators aim to answer the above questions through the following primary and secondary outcomes:

Primary outcomes Is there a difference in pain scores reported by the patient at 24 hours following LA-TAP versus no TAP block? Is there a clinically significant difference in cumulative postoperative opioid consumption, expressed as milligram morphine equivalents (MMEs) at 24 hours following LA-TAP blocks versus no TAP block? Secondary outcomes Is there a difference between study groups in pain scores at 48 & 72 hours? Is there a difference between study groups in total opioid consumption (MMEs) by 48 & 72 hours? Is there a difference between the study groups for reported post-operative nausea and vomiting? Is there a difference between the study groups in operating time? Is there a difference between the study groups in the length of Hospital stay? Is there a difference between the study groups in patient's satisfaction?

DETAILED DESCRIPTION:
Investigators aim to answer the above questions through the following primary and secondary outcomes:

Primary outcomes Is there a difference in pain scores reported by the patient at 24 hours following LA-TAP versus no TAP block? Is there a clinically significant difference in cumulative postoperative opioid consumption, expressed as milligram morphine equivalents (MMEs) at 24 hours following LA-TAP blocks versus no TAP block? Secondary outcomes Is there a difference between study groups in pain scores at 48 & 72 hours? Is there a difference between study groups in total opioid consumption (MMEs) by 48 & 72 hours? Is there a difference between the study groups for reported post-operative nausea and vomiting? Is there a difference between the study groups in operating time? Is there a difference between the study groups in the length of Hospital stay? Is there a difference between the study groups in patient's satisfaction?

Patients will be randomized in two arms , LA-TAP , NO-TAP block . Each patient would fill out the pain score sheet and number of narcotic medications she used in first 24h, 48h and 72 h post operatively .

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old and above
* English speaking
* patients with capacity to consent
* Elective laparoscopic and robotic benign genecology cases
* Elective laparoscopy/ robotic hysterectomy
* Elective laparoscopy/robotic myomectomy
* ERAS (enhanced recovery after surgery) protocol applied

Exclusion Criteria:

* Pregnant women
* patients with positive urine pregnancy test in pre operative
* emergency procedures
* Procedure requiring staging or debulking
* surgeries that convert to laparotomy
* patients with allergy to local/systemic anaesthesia or analgesia
* Inability to undergo normal anesthesia induction process
* ASA III or higher
* history of pain relief medication dependence
* history of substance abuse
* end stage chronic kidney disease
* advanced liver disease
* history of chronic pain
* history of taking opioids or neuropathic agents regularly prior to surgery
* BMI of 50 or over
* skin infections at the site of TAP block injection or port sites.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
pain scores at 24 hours in LA-TAP and NO TAP block groups | 24 hour post op
  numeric pain score (NPS)pain scores at 24 hours will include the average pain score at rest reported by the patient in the first 24 hours.
Amount and type of opioid consumption , based on Questionnaire's information . between LA-TAP , UG-TAP and No TAP groups at 24 hours post operatively | 24 hour post op
  MME will be calculated as the cumulative amount of opioid intake in the 24 hours following anesthesia end time.

SECONDARY OUTCOMES:
Numeric pain score (NPS) based on questionnaire's information at 48 hours & 72 hours post operatively , in LA-TAP , UG-TAp and no TAP groups | 48 -72 hour post operative
  numeric pain score (NPS)
amount of narcotic , per milligram and type of opiod consumption at 48 & 72 hours post operatively ? | 48 -72 hours post operative
  morphine equivalent dose of narcotic use
Nausea and vomiting post operatively , based on questionnaire's information at first 72 h post op | first 72 hours post operative
  nausea and vomiting, yes or no .

CONTACTS AND LOCATIONS:
Overall Officials: Farinaz Seifi, MD, FACOG, Principal Investigator — Yale University Obstetrics, Gynecology & Reproductive Sciences
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No